CLINICAL TRIAL: NCT03357003
Title: Observational Study (and Blood Samples Without Genetics Analysis) Tramadol Clinical Efficiency and Tolerance Correlated to O-desmethyltramadol/Tramadol Ratio (CLINCYTRAM)
Brief Title: Tramadol Clinical Efficiency and Tolerance Correlated to O-desmethyltramadol/Tramadol Ratio (CLINCYTRAM)
Acronym: CLINCYTRAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: CaenUH
Record Dates: First submitted 2017-03-07; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Observational study — Comparison between O-desmethyltramadol/tramadol ratio and tramadol clinical efficiency and tolerance

SUMMARY:
Tramadol is a grade II analgesics as World Health Organization definition. It can both be an agonist on mu receptors, which provides it a low opioid action, and also be a Serotonin-norepinephrine reuptake inhibitor, which act on neuropathic pain.

Tramadol is metabolized by P450 2D6 cytochrome (CYP2D6) in O-desmethyltramadol (O-dt) which is the most active form on the pharmacologic side (analgesic effect 2 to 4 times more powerful than tramadol itself).

In caucasian population, 5 to 10% of patients are genetically qualified as "poor metabolizer phenotype"; this status is correlated to a lower analgesic efficiency compared to "rapid metabolizer".

A multicenter study, CYTRAM, is under publication and allowed measurement of blood ratio O-dT/tramadol as a way to know the phenotype of CYP2D6 to detect "poor metabolizer phenotype" status.

Indeed, blood ratio O-dT/tramadol threshold under 0.1 detects " poor metabolizer phenotype " status for postoperative patients treated by tramadol, with a good sensibility (87,5%) and specificity (83.8%).

Which impacts for current practice? The next step is to know if this blood ratio is linked to an analgesic efficiency and a good tolerance for tramadol. A "poor metabolizer phenotype" patient would have no benefit of tramadol posology increasing. Therefore, phenotype detection, thank to blood ratio, could allow to switch quickly tramadol to another analgesic treatment for "poor metabolizer phenotype" patients.

The main objective of the study is to forge a link between O-dT/tramadol ratio and analgesic efficiency. Secondary objectives investigate side effects and frequency related to O-dT/tramadol ratio and pain relief, and also impact of CYP2D6 - inhibitor treatments on the blood ratio.

If there is a correlation between this blood ratio and treatment efficiency and tolerance, O-dT/tramadol ratio's detection will allow a better adaptation for some treatments metabolized by CYP2D6. Therefore, this evolution will contribute to health quality and health safety improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old treated by tramadol for at least 48h
* Tramadol posology between 100 and 400 mg/d (oral treatment) and until 600 mg/d (veinous treatment), recommended dosage
* Patients with nociceptive pain, definite etiology, combined or not with neuropathic pain
* Caucasian patient
* Patient able to give his/her informed consent
* Patient able to estimate himself/herself pain with pain scale for at least 48h

Exclusion Criteria:

* Age < 18 years old
* Patient with chronic pain (>3 month) or not definite
* Tramadol posology >400 mg/d (oral treatment) or > 600 mg/d (veinous treatment)
* Patients with absolute Tramadol contraindication
* Chronic endstage kidney failure antecedent (Cl cockcroft < 10mL/min) and liver failue antecedent
* Concomitant analgesic treatment, except paracetamol or stopped less than 48h ago
* Pregnant or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from nociceptive pain, combined or not with neuropathic pain, requiring tramadol treatment, grade II analgesics (WHO)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Ratio measurement : O-desmethyltramadol blood concentration/ tramadol blood concentration | at 48 hours
visual analogic pain scale (1 to 10) | at 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France